CLINICAL TRIAL: NCT05022082
Title: Comparison of the Efficiency of Chest Physiotherapy Applied in a Different Order in Pediatric Intensive Care Patients
Brief Title: The Efficiency of Chest Physiotherapy Applied in a Different Order
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Selmin Kose (Other)
Responsible Party: Sponsor-Investigator, Selmin Kose, Assistant Professor, Biruni University
Organization: Biruni University (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: BIRUNIUNIVERSITY
Record Dates: First submitted 2021-07-29; First posted 2021-08-26 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Respiratory Disease
Keywords: chest physiotherapy; aspiration; inhaler drugs; child; nurse
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Masking Description: The researchers (are nurses) have roles of care provider and also investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chest Physiotherapy- Aspiration- Inhaler drugs group (Experimental): The study group (n=21) will first receive chest physiotherapy (tapotement or vibration) and aspiration, followed by inhaler drug therapy.
  Interventions: Other: Chest Physiotherapy- Aspiration- Inhaler drugs group
- Inhaler drugs- Chest Physiotherapy- Aspiration group (Other): The control group (n=21) will be administered the inhaler drug routinely administered in the intensive care unit where the study is conducted and then receive chest physiotherapy (tapotement or vibration), then nasopharyngeal and oropharyngeal aspiration
  Interventions: Other: Chest Physiotherapy- Aspiration- Inhaler drugs group

INTERVENTIONS:
Other: Chest Physiotherapy- Aspiration- Inhaler drugs group — In the intensive care unit where the study was conducted, the patients who have a respiratory disorder and receive supplemental oxygen therapy with non-invasive mechanical ventilation or an oxygen mask are first administered an inhaler drug therapy placed in the physician's order. It is followed by chest physiotherapy and then oropharyngeal and nasopharyngeal aspiration. However, in practice rendered by the researcher, it is suggested that when chest physiotherapy and aspiration are administered in the first place and then followed by an inhaler drug therapy, it might have a more positive impact on the patient's physiologic parameters.

SUMMARY:
This study intends to compare the impact of chest physiotherapy applied with two different methods on physiologic parameters in children hospitalized in the intensive care unit. In the intensive care unit where the study was conducted, the patients who have a respiratory disorder and receive supplemental oxygen therapy with non-invasive mechanical ventilation or an oxygen mask are first administered an inhaler drug therapy placed in the physician's order. It is followed by chest physiotherapy and then oropharyngeal and nasopharyngeal aspiration. However, in practice rendered by the researcher, it is suggested that when chest physiotherapy and aspiration are administered in the first place and then followed by an inhaler drug therapy, it might have a more positive impact on the patient's physiologic parameters. For this reason, it is intended to compare the efficiency of chest physiotherapy applied in a different order.

DETAILED DESCRIPTION:
42 children who complied with the inclusion criteria will be included in the study. The mother or father of the children hospitalized in the pediatric intensive care unit of the hospital where the study is conducted will be given information about the study and asked to sign the "Informed Voluntary Consent Form". After the family's approval, they will be asked to fill out the "Parent Introductory Information Form".

The randomization method will be used to create the control group and the study group. Children to be included in the study will be placed in the groups with the randomized controlled method with 21 children in each group. The randomization of the study will be made with the online program available at the URL address https://www.randomizer.org/. Before entering the sample size in the program, lots will be drawn, and the 1st set will be assigned to the control group, and the 2nd set will be assigned to the study group. In order to determine in which group the children involved in the study will be placed, numbers from 1 to 42 will be entered into the program without repetition. Children that will constitute the study group through the program will be randomly distributed into 2 groups.

The control group (n=21) will be administered the inhaler drug routinely administered in the intensive care unit where the study is conducted and then receive chest physiotherapy (tapotement or vibration), then nasopharyngeal and oropharyngeal aspiration. The study group (n=21) will first receive chest physiotherapy (tapotement or vibration) and aspiration, followed by inhaler drug therapy.

The "Patient Data Collection Forms" of both groups will be filled out. Chest physiotherapy will follow the "Tapotement and Vibration Application Procedure," and aspiration will follow the "Nasopharyngeal and Oropharyngeal Aspiration Application Procedure". The "Patient Physiologic Parameter Assessment Form" information will be recorded before the application and 30 minutes after the application. It is known that the stress hormones epinephrine and norepinephrine half-life is 1-3 minutes, and it is believed that after a stressful invasive intervention, the release of stress hormones increases but turns back to their normal levels in 15-20 minutes (Puntillo et al. 2001). Based on this information, vital findings will be recorded in the "Patient Physiologic Parameter Assessment Form" after 30 minutes.

Obtained data will be evaluated using necessary statistical tests in the computer environment. Evaluation methods will be selected considering if data is distributed homogenously. If it has a homogenous distribution, parametric tests will be used. If it does not have a homogenous distribution, non-parametric methods will be used.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized patients at Cerrahpaşa Faculty of Medicine Pediatric Intensive Care Unit 1,
* Aged between 1 months-6 years,
* Having been in intensive care for at least two days,
* Concious pediatric patient,
* Receiving supplemental oxygen therapy with non-invasive mechanical ventilation or an oxygen mask,
* Being administered chest physiotherapy (Tapotement or Vibration),
* Being administered oropharyngeal and nasopharyngeal aspiration,
* Inhaler drug therapy included in the patient's order,
* Parents, volunteering for the study.

Exclusion Criteria:

* Parents not volunteering for the study,
* Patients younger than 1-month or older than 6-years old,
* Not receiving supplemental oxygen therapy with non-invasive mechanical ventilation or an oxygen mask
* Not being administered oropharyngeal and nasopharyngeal aspiration,
* Inhaler drug therapy is not included in the physician's order.

Ages: 1 Month to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 42 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Physiological Parameter Assessment Form Showing The Change In Heart Rate | This procedure will be applied to each patient for 30 minutes 4 times a day. It will be applied for at least 2 days and until the patient is discharged.
  Chest physiotherapy applied in a different order in pediatric intensive care patients causes a difference in the patient's physiologic parameters.This form prepared by the researcher includes recording pulse rate/min in the clinic. The researcher will be assessed the pulse/min at least four times before and after the chest physiotherapy in a day. The "Patient Physiologic Parameter Assessment Form" information will be recorded before the application and 20 minutes after the application. It is known that the stress hormones epinephrine and norepinephrine half-life is 1-3 minutes, and it is believed that after a stressful invasive intervention, the release of stress hormones increases but turns back to their normal levels in 15-20 minutes. Based on this information, the pulse will be recorded in the "Patient Physiologic Parameter Assessment Form" after 20 minutes.

SECONDARY OUTCOMES:
Physiological Parameter Assessment Form Showing The Change In SPO2% | This procedure will be applied to each patient for 30 minutes 4 times a day. It will be applied for at least 2 days and until the patient is discharged.
  Chest physiotherapy applied in a different order in pediatric intensive care patients causes a difference in the patient's physiologic parameters.This form prepared by the researcher includes recording SPO2% in the clinic. The researcher will be assessed the SPO2% at least four times before and after the chest physiotherapy in a day. The "Patient Physiologic Parameter Assessment Form" information will be recorded before the application and 30 minutes after the application. It is known that the stress hormones epinephrine and norepinephrine half-life is 1-3 minutes, and it is believed that after a stressful invasive intervention, the release of stress hormones increases but turns back to their normal levels in 15-20 minutes. Based on this information, the SPO2% will be recorded in the "Patient Physiologic Parameter Assessment Form" after 30 minutes.

OTHER OUTCOMES:
Physiological Parameter Assessment Form Showing The Change In Respiration rate/min | This procedure will be applied to each patient for 30 minutes 4 times a day. It will be applied for at least 2 days and until the patient is discharged.
  Chest physiotherapy applied in a different order in pediatric intensive care patients causes a difference in the patient's physiologic parameters.This form prepared by the researcher includes recording respiration rate/min in the clinic. The researcher will be assessed the respiration rate/min at least four times before and after the chest physiotherapy in a day. The "Patient Physiologic Parameter Assessment Form" information will be recorded before the application and 30 minutes after the application. It is known that the stress hormones epinephrine and norepinephrine half-life is 1-3 minutes, and it is believed that after a stressful invasive intervention, the release of stress hormones increases but turns back to their normal levels in 15-20 minutes. Based on this information, the respiration rate/min will be recorded in the "Patient Physiologic Parameter Assessment Form" after 30 minutes.
Physiological Parameter Assessment Form Showing The Change In Blood pressure (mmHg) | This procedure will be applied to each patient for 30 minutes 4 times a day. It will be applied for at least 2 days and until the patient is discharged.
  Chest physiotherapy applied in a different order in pediatric intensive care patients causes a difference in the patient's physiologic parameters.This form prepared by the researcher includes recording respiration blood pressure (mmHg) in the clinic. The researcher will be assessed the blood pressure (mmHg) at least four times before and after the chest physiotherapy in a day. The "Patient Physiologic Parameter Assessment Form" information will be recorded before the application and 30 minutes after the application. It is known that the stress hormones epinephrine and norepinephrine half-life is 1-3 minutes, and it is believed that after a stressful invasive intervention, the release of stress hormones increases but turns back to their normal levels in 15-20 minutes. Based on this information, the blood pressure (mmHg) will be recorded in the "Patient Physiologic Parameter Assessment Form" after 30 minutes.
Physiologic Parameter Assessment Form Showing The Change In Blood gas (mmHg) | The blood gas will driven twice a day routinely.
  In the clinic, although the time varies depending on the physician's request, the blood gas will driven twice a day routinely.

CONTACTS AND LOCATIONS:
Overall Officials: SEVVAL UNAL, RN, Principal Investigator — Istanbul University-Cerrahpaşa Cerrahpaşa School of Medicine
Locations (1):
- Selmin Köse, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Due to Hospital policy, the individual participant data can not be shared with anyone except researchers.